CLINICAL TRIAL: NCT04107935
Title: Telemedicine for Reach, Education, Access and Treatment-ongoing
Acronym: TREAT-ON
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to COVID-19 pandemic, we were unable to meet our recruitment goal during the grant period.
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Linda Siminerio, Professor, University of Pittsburgh
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY19080005; 1R34DK123370-01 (NIH)
Record Dates: First submitted 2019-09-25; First posted 2019-09-27 (Actual); Results first posted 2023-11-18 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Diabetes Mellitus
Keywords: Self management education and support; Telemedicine; Rural
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental)
  Interventions: Behavioral: TREAT-ON
- Usual Care (Other)
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: TREAT-ON — TREAT-ON is a DE-driven self-management and support program that is delivered primarily through a real-time telemedicine videoconferencing platform. Like the usual care intervention, "high risk" patients with DM receiving care in underserved practices will be identified by a nurse practice-based manager (PCBM) and referred to a DE for self management services. Participants will complete an initial face-to-face visit with the DE to assess needs and develop a self-management treatment plan and goals. Via telemedicine videoconferencing, follow-up visits will be delivered by the DE to participants in their homes. Follow-up visits will be used to evaluate and support progress towards meeting and sustaining self-management goals and outcomes.
  Arms: Intervention
Behavioral: Usual Care — A retrospective control group will be formed from individuals who have previously participated in a program called the "Diabetes High Risk Initiative." In this program, patients receiving care in underserved practices are identified by a nurse PBCM to be at high risk for DM complications and/or unplanned care and referred to a DE for self management services delivered through primary care. Patients typically participate in one face-to-face visit with the DE to assess needs and develop self-management goals and then one to two follow-up encounters (generally conducted by telephone) with the PBCM or DE.
  Arms: Usual Care

SUMMARY:
Diabetes (DM) management requires health care providers to provide patients with the appropriate amount of time, education and support that are necessary for quality care. Unfortunately, this is often impeded by limited access to resources, particularly in rural communities where DM rates are high and providers are scarce. Therefore, study investigators propose addressing these issues by implementing a model of care that includes diabetes educator (DE)-led planned visits with a real-time videoconferencing telemedicine program for ongoing patient support to improve DM outcomes.

DETAILED DESCRIPTION:
Health care systems need to seek ways through quality improvement, care coordination, and workforce capacity to support quality care. It has been proposed that new models of care coupled with technology are needed. DM provides an ideal model for testing new approaches as the number of people with DM continues to rise, with an inverse shortage of health providers available to meet their needs. Most patients with Type 2 DM (T2DM) are seen in primary care (PC) where providers report barriers to comprehensive care that include limited time, educational resources, added workload and feeling ill-equipped to counsel patients on behavior change. Efforts to restructure PC are underway, like DE-led planned management visits, reported to improve healthy behaviors and outcomes in patients at high risk. DEs are well suited to support the skills, decision making, self-care behaviors, problem solving and active collaboration with the care team that serve as the foundation for diabetes self-management education and key to an effective planned visit. DEs supporting care and self-management education in PC have been shown to improve access and outcomes. For patients to sustain a lifetime of behavior to effectively self-manage, continued support to sustain the ongoing skills, knowledge, and behaviors required to manage their condition is needed. Given the need for enduring support and scarcity of providers, particularly in underserved rural areas, efforts to understand how best to re-design practice to involve DEs in PC and utilize technology to enable and scale engagement in self-management and ongoing support must be considered. The purpose of this application is to evaluate the deployment of Telemedicine for Reach, Education, Access, Treatment and Ongoing Support (TREAT-ON), a DE-driven, PC-based telemedicine model that relies on PC practice redesign to afford access to real-time ongoing support. Investigators hypothesize that the TREAT-ON model will help individuals identified as being high risk in an underserved rural community to achieve and sustain improvements in clinical, psychosocial and behavioral outcomes, and aim to demonstrate the model's viability in terms of feasibility and acceptability to inform future testing of TREAT-ON.

ELIGIBILITY:
Inclusion Criteria:

* Intervention group: UPMC Health Plan patient-members who are 18-75y, have diagnosis of type 2 diabetes, are considered "high risk" (HbA1c >9%), receiving care at participating Federally Qualified Health Centers, and willing and able to participate in a technology-supported intervention.
* Control group: The control group will be selected from individuals who have already participated in the UPMC Health Plan's Diabetes High Risk Initiative.

Exclusion Criteria:

* Non UPMC Health Plan patients
* Not enrolled in the UPMC Health Plan Diabetes High Risk Initiative
* Less than 18 or greater than 75 years of age
* Unwilling/unable to participate in the telemedicine diabetes education program

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2020-02-04 (Actual); Primary Completion 2022-08-04 (Actual); Study Completion 2022-12-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda Siminerio, RN, PhD, CDE, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
After completion of the study, study investigators will prepare a consolidated dataset with all data collected as part of this study (e.g., clinical, behavioral, psychosocial, and satisfaction). All potentially identifying information will be removed. In addition, study investigators will prepare a Manual of Operations with a detailed description of the diabetes self-management and support intervention, the technology delivery system and a full description of the TREAT-ON model for dissemination.
Supporting Information: Study Protocol, ICF
Time Frame: Study protocol and data set - After publication. ICF - After data collection is completed.
Access Criteria: Study protocol and data set - other researchers will have to request access. ICF will be added to clinicaltrials.gov protocol

REFERENCES:
- [Derived] Siminerio L, Krall J, Johnson P, Ruppert K, Hammoudeh R, Bandi A, Ng JM. Examining a Diabetes Self-Management Education and Support Telemedicine Model With High-Risk Patients in a Rural Community. J Diabetes Sci Technol. 2023 Sep;17(5):1190-1197. doi: 10.1177/19322968231180884. Epub 2023 Jun 20. PMID 37338130

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from federally qualified health centers that offered a diabetes program to high risk patients who met certain criteria.
Pre-assignment Details: Usual care is a historical comparison group, therefore usual care participants were not considered to be enrolled into the study.
Groups:
- Intervention: Intervention: TREAT-ON is a DE-driven self-management and support program that is delivered primarily through a real-time telemedicine videoconferencing platform. Like the usual care intervention, "high risk" patients with DM receiving care in underserved practices will be identified by a nurse practice-based manager (PCBM) and referred to a DE for self management services. Participants will complete an initial visit with the DE to assess needs and develop a self-management treatment plan and goals. Via telemedicine videoconferencing, follow-up visits will be delivered by the DE to participants in their homes. Follow-up visits will be used to evaluate and support progress towards meeting and sustaining self-management goals and outcomes.
- Usual Care: Usual Care: A retrospective control group will be formed from individuals who have previously participated in a program called the "Diabetes High Risk Initiative." In this program, patients receiving care in underserved practices are identified by a nurse PBCM to be at high risk for DM complications and/or unplanned care and referred to a DE for self management services delivered through primary care. Patients typically participate in face-to-face visit(s) with the DE to assess needs and develop self-management goals and then one to two follow-up encounters (generally conducted by telephone) with the PBCM or DE.
Period: Overall Study
Arm/Group | Intervention | Usual Care
Started | 43 | 30
Completed | 42 | 30
Not Completed | 1 | 0
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Population: Usual care participants were identified through retrospective chart review; they were not formally enrolled in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Usual Care | Total
Number analyzed (Participants) | 43 | 30 | 73
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 41 | 27 | 68
  >=65 years | 2 | 3 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 19 | 43
  Male | 19 | 11 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 41 | 30 | 71
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 5 | 13
  White | 35 | 25 | 60
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 43 | 30 | 73
Hemoglobin A1c [Mean (Inter-Quartile Range); unit: % glycated hemoglobin] | 10.8 [9.9 to 12.5] | 10.4 [9.8 to 11.8] | 10.6 [9.8 to 12.2]

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Glycemic Control
Description: Average change in HbA1c every 3 months from baseline through 12 months was assessed using mixed model regression with repeat measures and therefore there is only one result reported per arm.
Time Frame: Change every 3 months for 12 months.
Population: Using propensity score matching, 30 intervention participants were paired with 30 usual care participants to compare changes in hemoglobin A1c.
Measure: Mean (95% Confidence Interval); unit: % change
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 30 | 30
% change | -0.14 [-0.2017 to -0.0761] | -0.14 [-0.2046 to -0.0712]
Statistical Analysis 1: Comparison: Intervention vs Usual Care; Test type: Superiority; p = 0.9830, Mixed Models Analysis — Propensity score matching was used to form pairs of intervention and control participants. Specifically, a greedy matching procedure with a matching caliper of 0.2 of the standard deviation of the logit of the propensity score was used; Since baseline characteristics achieved a good balance, those variables were not entered into the propensity score matched model

2. Secondary Outcome: Change From Baseline in Diabetes Self-care Behavior [Diet] Across 3 Month Intervals for 12 Months.
Description: Summary of Diabetes Self-care Activities Measure was used to evaluate self-care with questions about number of days in a week that the participant reports self-care behaviors. Individual items are scored 0 (minimum) to 7 (maximum) for number of days the behavior is performed. The total possible score ranges from 0 to 7. The higher the score for dietary behavior, the better. For this study, average change in scores from baseline through 12 months was assessed using mixed model regression with repeat measures and therefore there is only one result reported per arm.
Time Frame: Change every 3 months for 12 months total.
Population: Intervention participants
Measure: Mean (95% Confidence Interval); unit: Score on a scale
Groups:
- Intervention Self-management Goal Achievers: Participants in the intervention group who achieved their diabetes self-management goal(s). These are goals set to improve one or more self-care behavior(s) salient to diabetes management (e.g., healthy eating, exercise, coping, taking medication, monitoring, reducing risks and problem solving).
- Intervention Self-management Goal NON-achievers: Participants in the intervention who did not achieve their self-management goal(s). These are goals set to improve one or more self-care behavior(s) salient to diabetes management (e.g., healthy eating, exercise, coping, taking medication, monitoring, reducing risks and problem solving).
Arm/Group | Intervention Self-management Goal Achievers | Intervention Self-management Goal NON-achievers
Number analyzed (Participants) | 27 | 15
Score on a scale | 0.08 [0.0006 to 0.1563] | 0.09 [-0.02313 to 0.2092]
Statistical Analysis 1: Comparison: Intervention Self-management Goal Achievers vs Intervention Self-management Goal NON-achievers; Test type: Superiority; p = 0.8365, Mixed Models Analysis — Adjusted for age, race, body mass index, and time

3. Secondary Outcome: Change From Baseline in Diabetes Distress Across 3 Month Intervals for 12 Months
Description: Diabetes distress was evaluated with the 17-item Diabetes Distress Scale, which assesses four dimensions of distress - emotional, regimen, interpersonal and physician (Polonsky et al, 2005), and has shown a consistent pattern of relationships with HbA1c, diabetes self-efficacy, diet and physical activity in multiple samples of patients with T2DM (Fisher et al, 2012). Individual items are scored from 1 to 6; total scores are the average of all individual item scores; higher scores indicate greater distress (represents worse outcome). Possible score range 1 to 6. For this study, average change in scores every 3 months from baseline through 12 months was assessed using mixed model regression with repeat measures and therefore there is only 1 result reported per arm.
Time Frame: Change every three months for 12 months total
Population: Participants in the intervention group
Measure: Mean (95% Confidence Interval); unit: Score on scale
Arm/Group | Intervention Self-management Goal Achievers | Intervention Self-management Goal NON-achievers
Number analyzed (Participants) | 27 | 15
Score on scale | 0.1693 [-0.2060 to 0.5446] | -0.01655 [-0.5543 to 0.5212]
Statistical Analysis 1: Comparison: Intervention Self-management Goal Achievers vs Intervention Self-management Goal NON-achievers; Test type: Superiority; p = 0.5727, Mixed Models Analysis — Adjusted for age, race, body mass index, and time

4. Secondary Outcome: Change From Baseline in Diabetes Empowerment Across 3 Month Intervals for 12 Months
Description: Empowerment was measured using the 8-item Diabetes Empowerment Scale-Short Form, which measures an individual's perceived ability to manage psychosocial aspects of diabetes, assess dissatisfaction and readiness to change self-management plans and set and achieve diabetes goals (Anderson et al, 2000; Anderson et al, 2003). Possible scores are 1 to 5 for each item, summed for a possible total score of 8 to 40. Higher scores indicate greater empowerment (better outcome). For this study, average change in scores every 3 months from baseline through 12 months was assessed using mixed model regression with repeat measures and therefore there is only 1 result reported per arm.
Time Frame: Change every 3 months for 12 months total
Population: Participants in the intervention group
Measure: Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Intervention Self-management Goal Achievers | Intervention Self-management Goal NON-achievers
Number analyzed (Participants) | 27 | 15
Score on a scale | 0.01418 [-0.02730 to 0.05565] | 0.01129 [-0.04932 to 0.07189]
Statistical Analysis 1: Comparison: Intervention Self-management Goal Achievers vs Intervention Self-management Goal NON-achievers; Test type: Superiority; p = 0.9381, Mixed Models Analysis — Adjusted for age, race, body mass index, and time

5. Secondary Outcome: Intervention Acceptability
Description: Telemedicine Usability Questionnaire was used to assess telehealth usefulness, ease of use and learnability, interface quality, patient-clinician interaction, reliability, satisfaction and future use and included additional items specific to this study. Individual items are scored on a scale from one to five, with one being strongly disagree to five being strongly agree. Scores are averaged for a possible score range of one to five. The higher the score infers the better the usability of the telehealth service.
Time Frame: 12 months
Population: Participants in intervention group who completed the survey
Measure: Mean (Inter-Quartile Range); unit: Score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 38
Score on a scale | 4.6 [3.95 to 5]

6. Secondary Outcome: Change From Baseline in Medication Adherence Across 3 Month Intervals for 12 Months
Description: Medication adherence was assessed with the 8-item Morisky Medication Adherence Scale (MMAS-8). The scales includes 8 items. Scores can range from 0 to 8; the higher the score, the more adherent the respondent is considered. For this study, average change in scores every 3 months from baseline through 12 months was assessed using mixed model regression with repeat measures and therefore there is only 1 result reported per arm.
Time Frame: Change every 3 months for 12 months total
Population: Participant in the intervention
Measure: Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Intervention Self-management Goal Achievers | Intervention Self-management Goal NON-achievers
Number analyzed (Participants) | 27 | 15
Score on a scale | 0.1419 [0.06095 to 0.2229] | 0.1044 [-0.01793 to 0.2267]
Statistical Analysis 1: Comparison: Intervention Self-management Goal Achievers vs Intervention Self-management Goal NON-achievers; Test type: Superiority; p = 0.608, Mixed Models Analysis — Adjusted for age, race, body mass index, and time

ADVERSE EVENTS:
Time Frame: 12 months
Description: Usual care group was a historical comparison group.
Arm/Group | Intervention | Usual Care
All-Cause Mortality (participants affected / at risk) | 1/43 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/30
Other Adverse Events (participants affected / at risk) | 0/43 | 0/30

LIMITATIONS AND CAVEATS:
The trial was implemented when the COVID-19 pandemic started and there were restrictions and challenges with meeting in person to enroll patients. Also, the study design included a historic control group to make best use of available resources, but propensity score matching only matched 30 participant control/intervention pairs. Furthermore, a retrospective versus parallel control group design prevented collecting behavioral psychosocial and satisfaction data for the control group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2023-07-24): https://cdn.clinicaltrials.gov/large-docs/35/NCT04107935/Prot_001.pdf
  • Statistical Analysis Plan (2023-07-24): https://cdn.clinicaltrials.gov/large-docs/35/NCT04107935/SAP_002.pdf
  • Informed Consent Form (2020-08-05): https://cdn.clinicaltrials.gov/large-docs/35/NCT04107935/ICF_000.pdf